CLINICAL TRIAL: NCT01582178
Title: Warm Water Versus Room Temperature Water Immersion Colonoscopy - a Prospective, Randomized, Double-blind, Single-center Trial
Brief Title: Warm Water Versus Room Temperature Water Immersion Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitkovice Hospital (Other)
Responsible Party: Principal Investigator, Premysl Falt MD, Principal Investigator, Vitkovice Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: DDC VN 04
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Results first posted 2013-08-01 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Colorectal Cancer
Keywords: colonoscopy; warm water immersion; cool water immersion
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Warm Water Immersion Colonoscopy (Experimental): Colonoscopy using purely warm water (37°C) infusion during colonoscope insertion and room air insufflation during colonoscope withdrawal.
  Interventions: Procedure: Warm Water Immersion Colonoscopy
- Cool Water Immersion Colonoscopy (Active Comparator): Colonoscopy using purely room temperature water (20-24°C) infusion during colonoscope insertion and room air insufflation during colonoscope withdrawal.
  Interventions: Procedure: Cool Water Immersion Colonoscopy

INTERVENTIONS:
Procedure: Warm Water Immersion Colonoscopy — Colonoscopy using warm water (37°C) infusion for colonoscope insertion and room air insufflation during colonoscope withdrawal.
  Arms: Warm Water Immersion Colonoscopy
Procedure: Cool Water Immersion Colonoscopy — Colonoscopy using room temperature water (20-24°C) infusion for colonoscope insertion and room air insufflation during colonoscope withdrawal.
  Arms: Cool Water Immersion Colonoscopy

SUMMARY:
Water immersion insertion has been documented to decrease procedure-related discomfort during colonoscopy. There was used warm water infusion for colonoscope insertion in most of the water immersion colonoscopy trials.

The investigators have been using room temperature water (20-24°C) for water immersion and the investigators did not notice any drawback of it. In our opinion, it is simpler and cheaper option for water immersion colonoscopy and proof of its efficacy and safety could support the use of water immersion technique in routine practice.

The primary endpoint is cecal intubation time and the investigators suppose that the use of warm water infusion does not shorten it significantly. Patient comfort during colonoscope insertion, water consumption, length of the scope while reaching the cecum, need for external compression, need for positioning of the patient and endoscopist´s difficulty with colonoscopy will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

* outpatient diagnostic colonoscopy
* bowel prep with macrogolum
* initial 2 mg of midazolam i.v.
* signed informed consent form

Exclusion Criteria:

* planned therapeutic intervention
* colorectal surgery in history
* known inflammatory bowel disease or colorectal cancer
* refusal of sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Premysl Falt, MD, Principal Investigator — Digestive Diseases Center, Vitkovice Hospital
Locations (1):
- Digestive Diseases Center, Vitkovice Hospital, Ostrava, Czechia

REFERENCES:
- [Background] Falt P, Smajstrla V, Fojtik P, Tvrdik J, Urban O. Cool water vs warm water immersion for minimal sedation colonoscopy: a double-blind randomized trial. Colorectal Dis. 2013;15(10):e612-7. doi: 10.1111/codi.12336. PMID 23819909

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients older than 18 years referred to our unit for diagnostic outpatient colonoscopy. Subjects were excluded if they has a history of colorectal surgery, known diagnosis of IBD, chronic benzodiazepine use and if they refused sedation.
  The period between June and October 2012.
Pre-assignment Details: Subjects were not included if they did not fulfill inclusion criteria.
Period: Overall Study
Arm/Group | Warm Water Immersion Colonoscopy | Cool Water Immersion Colonoscopy
Started | 106 | 106
Completed | 100 | 101
Not Completed | 6 | 5
Not completed — Physician Decision | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Warm Water Immersion Colonoscopy | Cool Water Immersion Colonoscopy | Total
Number analyzed (Participants) | 106 | 106 | 212
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 43 | 90
  >=65 years | 59 | 63 | 122
Age Continuous [Mean (Standard Deviation); unit: years] | 61.2 (12.7) | 57.8 (14.2) | 59.5 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 49 | 97
  Male | 58 | 57 | 115
Region of Enrollment [Number; unit: participants]
  Czech Republic | 106 | 106 | 212

OUTCOME MEASURES:

1. Primary Outcome: Cecal Intubation Time
Time Frame: 3 months
Reporting Status: Not Posted

2. Secondary Outcome: Patient Comfort During Insertion Phase of the Colonoscopy
Time Frame: 3 months
Reporting Status: Not Posted

3. Primary Outcome: Cecal Intubation Time
Description: = time between introduction of the colonoscope into the anus and reaching the cecum.
Time Frame: 1-30
Measure: Mean (Standard Deviation); unit: minute
Arm/Group | Warm Water Immersion Colonoscopy | Cool Water Immersion Colonoscopy
Number analyzed (Participants) | 100 | 101
minute | 7.0 (3.4) | 6.9 (3.5)
Statistical Analysis 1: Comparison: Warm Water Immersion Colonoscopy vs Cool Water Immersion Colonoscopy; Test type: Superiority or Other; p = 0.89, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Warm Water Immersion Colonoscopy | Cool Water Immersion Colonoscopy
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/106
Other Adverse Events (participants affected / at risk) | 0/106 | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No